CLINICAL TRIAL: NCT04888884
Title: Loss of Independence (LOI) - a Rapid Alternative to Frailty Screening in a Swedish Emergency Department Setting
Brief Title: Loss of Independence - a Rapid Alternative to Frailty Screening in a Swedish ED Setting
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Daniel Wilhelms, Principal Investigator, University Hospital, Linkoeping
Other Study IDs: 2021-00875LOI
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Frailty; Frailty Syndrome; Emergency Department; Geriatric Assessment
MeSH Terms: conditions — Frailty; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study will investigate the correlation of a surrogate marker of frailty in relation to serious outcomes. Serious outcomes are defined as: mortality within 30 days, admission to hospital, length of stay in the Emergency Department (ED), in-hospital Length of Stay and revisits to the ED.

The exposure, frailty, will be assessed according to Loss of Independence (LOI) a possible low-cost quick tool to identify frailty in patients. The study population will be ED patients, >65 years of age in a Swedish regional health care system (Region Östergötland, Sweden), comprising three EDs in Linköping, Norrköping and Motala. The outcomes will be compared according to the degree of frailty and censored over 7, 30 and 90 days.

DETAILED DESCRIPTION:
Frailty is a common clinical syndrome in older adults that carries an increased risk for poor health outcomes including falls, incident disability, hospitalization and mortality.

The Loss of Independence (LOI) defined as inability to rise from a chair with or without existing aids, is a possible low cost surrogate marker to measure frailty. Several studies on triage scores for predicting mortality and need of hospital admission have identified LOI as one of the most important variables. LOI was prognostic in ED populations regarding mortality within 1-30 days in Denmark, Ireland and Tanzania. Data from the American College of Surgeons (ACS) National Surgical Quality Improvement Program (NSQIP) Geriatric Surgery Pilot Project showed that LOI was associated with higher rates of readmission and death after discharge in geriatric patients undergoing surgical procedures6.

The aim of this study will be to investigate if the frailty, as assessed with LOI, is associated with increased 30-day mortality in a Swedish ED context. Secondary outcomes include 7- and 90-day mortality, ED-length of stay, hospital admission, in-hospital length of stay, subsequent falls and medication changes. Additionally, we collect data on morbidity and comorbidities to assess the association with the level of frailty. Since this is a multicentre study, possible geographic differences will be studied as well. Based on the results of this study, possible interventions could be identified to improve the care of the frail geriatric patients presenting at the ED.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years
* able to answer questions to estimate frailty
* or have a proxy to answer questions

Exclusion Criteria:

* <65 years
* unable to answer questions to estimate frailty

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients of all gender at the age of ≥ 65 years seeking medical care at the three EDs in Region Östergötland.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality in 30 Days | All cause mortality up to 30 days from index visit
  Investigate level of mortality in cohort at 30 days

SECONDARY OUTCOMES:
Mortality in 7 and 90 days | All cause mortality up to 90 days from index visit
  Investigate level of mortality in cohort at 7 and 90 days
Admission to hospital | Hospital admission on index visit, censored at 90 days
  Investigate level of all cause admissions in cohort
ED length of stay | Length of stay at ED, censored at 4 days
  Investigate length of stay at ED
In-hospital length of stay | In-hospital length of stay from index visit, censored at 90 days
  Investigate in-hospital length of stay
Revisits to the ED | Number of newly registered visits to the ED after index visit, censored at 90 days
  Number of newly registered visits to the ED after index visit
Fall prevalence after index visit | Falls that resulted in further health care contacts after index visit, censored at 90 days
  Falls that resulted in further health care contacts
Alterations in medication during the visit | Alterations in medication during the ED visit and during the follow-up period, censored at 90 days
  Alterations in medication during the ED visit and during the follow-up period(based on codes for Anatomical, Therapeutic, Chemical classification (ATC-code)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Wilhelms, PhD, Principal Investigator — Linkoeping University
Locations (3):
- Sweden (3):
  - University Hospital Linköping, Linköping, Östergötland County
  - Medicinska Specialist Kliniken i Motala, Motala, Östergötland County
  - Vrinnevisjukhuset i Norrköping, Norrköping, Östergötland County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kellett J, Deane B. The Simple Clinical Score predicts mortality for 30 days after admission to an acute medical unit. QJM. 2006 Nov;99(11):771-81. doi: 10.1093/qjmed/hcl112. Epub 2006 Oct 17. PMID 17046859
- [Background] Kellett J, Deane B, Gleeson M. Derivation and validation of a score based on Hypotension, Oxygen saturation, low Temperature, ECG changes and Loss of independence (HOTEL) that predicts early mortality between 15 min and 24 h after admission to an acute medical unit. Resuscitation. 2008 Jul;78(1):52-8. doi: 10.1016/j.resuscitation.2008.02.011. Epub 2008 Apr 10. PMID 18406038
- [Background] Brabrand M, Folkestad L, Clausen NG, Knudsen T, Hallas J. Risk scoring systems for adults admitted to the emergency department: a systematic review. Scand J Trauma Resusc Emerg Med. 2010 Feb 11;18:8. doi: 10.1186/1757-7241-18-8. PMID 20146829
- [Background] Brabrand M, Lassen AT, Knudsen T, Hallas J. Seven-day mortality can be predicted in medical patients by blood pressure, age, respiratory rate, loss of independence, and peripheral oxygen saturation (the PARIS score): a prospective cohort study with external validation. PLoS One. 2015 Apr 13;10(4):e0122480. doi: 10.1371/journal.pone.0122480. eCollection 2015. PMID 25867881
- [Background] Rylance J, Baker T, Mushi E, Mashaga D. Use of an early warning score and ability to walk predicts mortality in medical patients admitted to hospitals in Tanzania. Trans R Soc Trop Med Hyg. 2009 Aug;103(8):790-4. doi: 10.1016/j.trstmh.2009.05.004. Epub 2009 Jun 21. PMID 19540542
- [Background] Berian JR, Mohanty S, Ko CY, Rosenthal RA, Robinson TN. Association of Loss of Independence With Readmission and Death After Discharge in Older Patients After Surgical Procedures. JAMA Surg. 2016 Sep 21;151(9):e161689. doi: 10.1001/jamasurg.2016.1689. Epub 2016 Sep 21. PMID 27409710